CLINICAL TRIAL: NCT04732000
Title: Oxidative Stress and Surgical Recovery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Martin Angst, Professor of Anesthesia, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 59401
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Results first posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Surgical Recovery; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetylcysteine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- N-acetyl cysteine (Active Comparator): N-acetyl cysteine will be administered as follows: A loading dose of 50 mg/kg will be started as a 1-hour infusion before surgical incision, and will be followed by a maintenance dose of 50 mg/kg administered over 4 hours.
  Interventions: Drug: N-acetyl cysteine
- Normal Saline (Placebo Comparator): Normal will be administered as follows: A normal saline infusion will administered at a rate and duration to mimic the N-acetyl cysteine administration.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: N-acetyl cysteine — Intravenous infusion started during the clinically indicated surgery at a rate of 50mg/kg over 1 hour followed by 50mg/kg over 3 hours. This will be an accumulated total of 100 mg/kg over 4 hours.
  Other Names: NAC
  Arms: N-acetyl cysteine
Other: Normal Saline — Intravenous infusion at a time and rate to mimic the active treatment. The infusion will be given over 4 hours beginning during the clinically indicated surgery
  Other Names: NS
  Arms: Normal Saline

SUMMARY:
Chronic pain, functional impairment and slow rates of recovery are key issues for patients after surgery and trauma. No preventative strategy in current use unequivocally modifies these rates, and few novel approaches have been tested. Furthermore, persistent postsurgical pain is a major route to chronic opioid use, opioid use disorder and, regrettably, opioid overdose. Most strategies designed to limit chronic pain or enhance functional recovery after surgery are directed at modulating peripheral and central nervous system activity and do not strongly modify the underlying tissue pathophysiology or fundamental systemic responses. Strategies limiting oxidative stress in the perioperative period, on the other hand, might limit tissue damage, organ dysfunction and immune system activation.

N-acetyl cysteine (NAC) is an antioxidant well-studied in the perioperative period; it is very safe, relatively inexpensive and widely available. The central hypothesis is, therefore, that perioperative administration of NAC will reduce perioperative oxidative stress, limit immune system activation and improve key indices of surgical recovery. Although the planned work will not comprehensively address this hypothesis, it will identify the most useful tools and help the researchers estimate the required sample sizes for more definitive externally funded efforts.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled interventional pilot study in 20 patients undergoing first-time total hip arthroplasty (THA) for chronic osteoarthritis at Stanford Medicine. The researchers will screen, enroll and collect biologic and behavioral data from 20 participants as outlined in previous observational and interventional clinical studies undertaken in close collaboration with the Department of Orthopedic Surgery. In particular, standard operating procedures for screening, recruiting, laboratory assessments, and clinical data collection are in place including eligibility screening via EPIC (EHR) ahead of patients' preoperative visit, coordinated recruitment and consenting during the pre-surgery visit including study- related laboratory work, further preoperative assessments after the visit (e.g. remote completion of questionnaires and direct import of results into REDCap), and real-time tracking of the data collection and storage process (e.g. including phone/email reminders if data are missing).

Repeated assessments of pain, physical function, and analgesic medication will be made before surgery, daily on postoperative days 1-3, and then twice a week in post-op weeks 1 - 6. Delirium will be measured days 1-3 while in-hospital. Additional data will include demographics (age, BMI, sex, race, and ethnicity), surgical/anesthesia data (e.g. duration), and medical/medication history.

Peripheral blood samples will be collected before surgery and 1hr and 24hr after surgery based on our prior study showing that monocyte activation (including STAT3, CREB and NFkB signaling responses in CD14+CD16- monocytes) early after surgery strongly correlates with delayed pain resolution and functional impairment. Exhaled breath samples will be collected intraoperatively prior to incision and at wound closure as well as at 1 and 24 hours after surgery.

N-Acetylcysteine infusion: A loading dose of 50 mg/kg will be started as a 1-hour infusion before surgical incision, and will be followed by a maintenance dose of 50 mg/kg administered over 4 hours. This is a standard dosing paradigm that is safe when used intraoperatively and rarely causes significant adverse effects (mainly allergic reactions).

Surgery and anesthesia: Participants will undergo unilateral hip arthroplasty performed by three surgeons using the same approach. The anesthetic and perioperative management of patients is standardized and follows ERAS-based recommendations.

Measures: Well-validated instruments will be used to assess pain, pain interference and function of the affected and operated joint including the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) adapted for patients undergoing lower extremity joint surgery, the Brief Pain Inventory (BPI) and the Surgical Recovery Scale (SRS). Opioid consumption will be quantified as intravenous hydromorphone equivalents (milligram/day) using widely accepted opioid conversion tables.

Sample analysis: Blood and plasma will be collected and processed for analysis with mass cytometry as previously described. A 39-parameter human CyTOF antibody panel will be applied that will allow the simultaneous analysis of 1) all major immune cell phenotypes 2) endogenous intracellular signaling responses (including the pSTAT3, pCREB and pNF-kB signal) and 3) intracellular markers of reactive aldehydes (i.e. 4-HNE and MDA signal).

Breath samples will be analyzed for aldehydes including formaldehyde, crotenaldehyde, and benzaldehyde using mass spectroscopy in the laboratory of Dr. Gross.

Plasma samples will be analyzed for free MDA and 4- HNE in baseline, 1 and 24-hour plasma samples in the laboratory of Dr. Clark.

Analysis and modeling of outcome data: Self-reported outcomes will be analyzed using the validated models associated with each outcome to extract a quantified and normalized number associated with recovery. The 60Htz actigraphy data will first be mined for patterns associated with daily activities (e.g. step counts) and intensity levels. Next, a baseline will be established using the data collected during and prior to surgery, for each variable. All variables will be normalized to this baseline to account for patient-specific effects. Finally, a multivariate linear model (with days passed since surgery as the response variable) will be used to model the entire actigraphy dataset. The area under the respective recovery curve of each patient according to this model will be used as an objective recovery outcome. In our preliminary studies (data not shown) this outcome has been found to be correlated with several aspects of the immune system.

Analysis and modeling of CyTOF data: The large number of data points (millions of cells per patient) and measured variables (tens of signaling pathways in hundreds of cell types) pose unique computational challenges that cannot be addressed using traditional bioinformatics tools. The researchers will develop a Bayesian framework that will combine a priori knowledge of the immune system with state-of-the-art mass cytometry profiling to build a predictive model of innate and adaptive immune cell signaling responses for each of the recovery outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18
2. Male of female
3. Planning to undergo primary total hip arthroplasty
4. Fluent in English
5. Willing and able to sign an informed consent form and HIPAA authorization and to comply with study procedures

Exclusion Criteria:

1. Infectious disease within the last month
2. Immune-suppressant therapy within the last 2 months (e.g., azathioprine or cyclosporine)
3. Chronic medication with potential immune-modulatory effects (e.g., daily oral morphine-equivalent intake > 30 mg)
4. Major surgery within the last 3 months or minor surgery within the last month.
5. History of substance abuse (e.g., alcoholism, drug dependency)
6. Pregnancy
7. Autoimmune disease interfering with data interpretation (e.g. lupus)
8. Renal, hepatic, cardiovascular, or respiratory diseases resulting in clinically relevant impaired function
9. Active malignancy
10. Participation in another clinical trial of an investigational drug or device within the last month that, in the investigator's opinion, would create an increased risk to the participant or compromise the integrity of the study
11. Other conditions compromising a participant's safety or the integrity of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin S Angst, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim DH, Pearson-Chauhan KM, McCarthy RJ, Buvanendran A. Predictive Factors for Developing Chronic Pain After Total Knee Arthroplasty. J Arthroplasty. 2018 Nov;33(11):3372-3378. doi: 10.1016/j.arth.2018.07.028. Epub 2018 Aug 4. PMID 30143334
- [Background] Zambelli VO, Gross ER, Chen CH, Gutierrez VP, Cury Y, Mochly-Rosen D. Aldehyde dehydrogenase-2 regulates nociception in rodent models of acute inflammatory pain. Sci Transl Med. 2014 Aug 27;6(251):251ra118. doi: 10.1126/scitranslmed.3009539. PMID 25163478
- [Background] Guo TZ, Wei T, Huang TT, Kingery WS, Clark JD. Oxidative Stress Contributes to Fracture/Cast-Induced Inflammation and Pain in a Rat Model of Complex Regional Pain Syndrome. J Pain. 2018 Oct;19(10):1147-1156. doi: 10.1016/j.jpain.2018.04.006. Epub 2018 Apr 30. PMID 29715519
- [Background] Gaudilliere B, Fragiadakis GK, Bruggner RV, Nicolau M, Finck R, Tingle M, Silva J, Ganio EA, Yeh CG, Maloney WJ, Huddleston JI, Goodman SB, Davis MM, Bendall SC, Fantl WJ, Angst MS, Nolan GP. Clinical recovery from surgery correlates with single-cell immune signatures. Sci Transl Med. 2014 Sep 24;6(255):255ra131. doi: 10.1126/scitranslmed.3009701. PMID 25253674
- [Background] Geiger-Maor A, Levi I, Even-Ram S, Smith Y, Bowdish DM, Nussbaum G, Rachmilewitz J. Cells exposed to sublethal oxidative stress selectively attract monocytes/macrophages via scavenger receptors and MyD88-mediated signaling. J Immunol. 2012 Feb 1;188(3):1234-44. doi: 10.4049/jimmunol.1101740. Epub 2012 Jan 4. PMID 22219328
- [Background] Aghaeepour N, Kin C, Ganio EA, Jensen KP, Gaudilliere DK, Tingle M, Tsai A, Lancero HL, Choisy B, McNeil LS, Okada R, Shelton AA, Nolan GP, Angst MS, Gaudilliere BL. Deep Immune Profiling of an Arginine-Enriched Nutritional Intervention in Patients Undergoing Surgery. J Immunol. 2017 Sep 15;199(6):2171-2180. doi: 10.4049/jimmunol.1700421. Epub 2017 Aug 9. PMID 28794234
- [Background] Fragiadakis GK, Gaudilliere B, Ganio EA, Aghaeepour N, Tingle M, Nolan GP, Angst MS. Patient-specific Immune States before Surgery Are Strong Correlates of Surgical Recovery. Anesthesiology. 2015 Dec;123(6):1241-55. doi: 10.1097/ALN.0000000000000887. PMID 26655308
- [Background] Pereira JEG, El Dib R, Braz LG, Escudero J, Hayes J, Johnston BC. N-acetylcysteine use among patients undergoing cardiac surgery: A systematic review and meta-analysis of randomized trials. PLoS One. 2019 May 9;14(5):e0213862. doi: 10.1371/journal.pone.0213862. eCollection 2019. PMID 31071081
- [Background] Kapstad H, Rokne B, Stavem K. Psychometric properties of the Brief Pain Inventory among patients with osteoarthritis undergoing total hip replacement surgery. Health Qual Life Outcomes. 2010 Dec 9;8:148. doi: 10.1186/1477-7525-8-148. PMID 21143926
- [Background] Baca Q, Marti F, Poblete B, Gaudilliere B, Aghaeepour N, Angst MS. Predicting Acute Pain After Surgery: A Multivariate Analysis. Ann Surg. 2021 Feb 1;273(2):289-298. doi: 10.1097/SLA.0000000000003400. PMID 31188202
- [Background] Aghaeepour N, Finak G; FlowCAP Consortium; DREAM Consortium; Hoos H, Mosmann TR, Brinkman R, Gottardo R, Scheuermann RH. Critical assessment of automated flow cytometry data analysis techniques. Nat Methods. 2013 Mar;10(3):228-38. doi: 10.1038/nmeth.2365. Epub 2013 Feb 10. PMID 23396282

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 participants signed consent, 24 were assigned to a study arm.
Groups:
- N-acetyl Cysteine: N-acetyl cysteine intravenous infusion started during the clinically indicated surgery at a rate of 50mg/kg over 1 hour followed by 50mg/kg over 3 hours to an accumulated total of 100 mg/kg over 4 hours.
- Normal Saline: Normal Saline intravenous infusion at a time and rate to mimic the active treatment given over 4 hours beginning during the clinically indicated surgery.
Period: Overall Study
Arm/Group | N-acetyl Cysteine | Normal Saline
Started | 13 | 11
Completed | 10 | 11
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Population: Participants who completed the protocol are included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | N-acetyl Cysteine | Normal Saline | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.0 [60.3 to 63.8] | 68.0 [61.0 to 74.0] | 64 [60 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 3 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 11 | 21
Body mass index [Median (Inter-Quartile Range); unit: kg/m2] | 27.7 [25.5 to 30.8] | 28.6 [26.4 to 33.5] | 28.3 [25.3 to 31.7]
Western Ontario & McMaster Universities Osteoarthritis Index - Pain [Median (Inter-Quartile Range); unit: score on a scale] — Score range: 0 (no pain) - 40 (worst pain)
  score on a scale | 24.5 [9.5 to 30.0] | 17.0 [15.0 to 29.0] | 22.0 [14.0 to 31.0]
Western Ontario & McMaster Universities Osteoarthritis Index - Function [Median (Inter-Quartile Range); unit: Score on a scale] — Score range: 0 (less physical function) - 68 (worst physical function)
  Score on a scale | 38.0 [18.5 to 43.8] | 32.0 [21.5 to 44.5] | 37.0 [20.0 to 44.0]
Opioids POD1 (IV Diluadid Eq.) [Median (Inter-Quartile Range); unit: mg/mL] | 3.4 [2.0 to 6.4] | 1.9 [0.9 to 5.6] | 2.3 [1.6 to 6.8]

OUTCOME MEASURES:

1. Primary Outcome: Phosphorylation of STAT-3 in MDSC (Myeloid-derived Suppressor Cells)
Description: STAT3 phosphorylation in MDSC cells is measured in all MDSC cells before (T0) and one day after surgery (T1) using mass cytometry. The median phosphorylation in this cell population is then determined for each time point. The change in phosphorylation is expressed as the arc sinh ratio of these two medians (ratio = arc sinh [median pSTAT3-T1/median pSTAT3-T0]).
Time Frame: Measurements will be made in samples collected before and 24 hours after surgery.
Population: Participants with samples that passes quality control were included in the analysis
Measure: Median (Inter-Quartile Range); unit: STAT3 archsinh ratio
Arm/Group | N-acetyl Cysteine | Normal Saline
Number analyzed (Participants) | 10 | 9
STAT3 archsinh ratio | 2.162 [1.966 to 2.264] | 2.025 [1.955 to 2.221]
Statistical Analysis 1: Comparison: N-acetyl Cysteine vs Normal Saline; Test type: Other; p = 0.5490, Mann Whitney test, 2-sided — The a priori threshold for statistical significance is < 0.05; Median Difference (Final Values) = -0.1373

2. Primary Outcome: Brief Pain Inventory Pain Score
Description: The Brief Pain Inventory was used to measure pain and pain interference following surgery. BPI Pain Composite Score was derived from worst pain, least pain, average pain, and pain right now subscale scores. BPI Pain Interference Composite Score (representing how pain interferes with daily life) was derived from general activity, mood, walking ability, normal work, relationships with others, sleep, and enjoyment of life subscale scores. Each composite score is the median value of the combined median values for each participant of the respective subscale scores (range for subscale and overall scores: 0 to 10, higher scores indicate more severe pain/pain interference).
Time Frame: post-operative week 6
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | N-acetyl Cysteine | Normal Saline
Number analyzed (Participants) | 10 | 11
score on a scale
  BPI Pain Composite Score | 1.3 [1.0 to 2.8] | 1.0 [0.3 to 1.3]
  BPI Pain Interference Composite Score | 2.5 [2.0 to 3.0] | 1.0 [0.0 to 1.0]

3. Secondary Outcome: Pain Score
Description: The Brief Pain Inventory will be used to measure pain following surgery at various time points. A composite score will be calculated 24 hours post op and will constitute the secondary end point. Overall score: median and interquartile range are reported across scores for worst pain, least pain, average pain, and right now pain. Pain interference score: represents how pain interferes with daily life. Score ranges: 0 to 10, higher scores indicate more severe pain.
Time Frame: Baseline through post-op day 1 (composite scores over 24 hours following surgery)
Population: Participants who completed the protocol are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | N-acetyl Cysteine | Normal Saline
Number analyzed (Participants) | 10 | 11
score on a scale
  Baseline - overall pain | 5.5 [2.1 to 7.1] | 4.5 [3.3 to 7.3]
  Post-op day 1 - overall pain | 4.3 [3.5 to 5.4] | 4.0 [2.5 to 6.5]
  Baseline - pain interference | 7.0 [5.3 to 7.8] | 5.0 [4.0 to 7.0]
  Post-op day 1 - pain interference | 6.5 [2.8 to 8.5] | 2.0 [2.0 to 5.5]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | N-acetyl Cysteine | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 6/13 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N-acetyl Cysteine (N=13) | Normal Saline (N=11)
Intestinal Cramps (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 1
Fever (≥37.2 C) (Investigations) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 0
Swelling of surgical leg and foot (Injury, poisoning and procedural complications) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Blisters above right hip (Infections and infestations) | 1 | 0
Chills (Investigations) | 0 | 1
Rash at site of regional anesthesia (Skin and subcutaneous tissue disorders) | 0 | 1
Full body rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hb ≤6.4 g/dL (Investigations) | 0 | 1
Shingles (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT04732000/Prot_000.pdf